CLINICAL TRIAL: NCT03701126
Title: Ultrasound Guided Transversus Abdominis Plane Block Versus Caudal Block in Inguinal Hernia Repair Surgery in Pediatrics
Brief Title: Ultrasound Guided TAP Block Versus Caudal Block in Pediatrics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohammed Abdullah Seliem Mekawy, Principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP/caudal block in pediatric
Record Dates: First submitted 2018-10-01; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): Transversus Abdominis Plane block using 1ml/kg of bupivacaine 0.25% under ultrasound guidance
  Interventions: Procedure: Transversus Abdominis Plane Block; Drug: Bupivacaine 0.25% Injectable Solution; Device: Ultra-sound guidance
- group B (Active Comparator): Caudal block using 1ml/kg of bupivacaine 0.25% under ultrasound guidance
  Interventions: Procedure: Caudal Block; Drug: Bupivacaine 0.25% Injectable Solution; Device: Ultra-sound guidance

INTERVENTIONS:
Procedure: Transversus Abdominis Plane Block — ultrasound (US) guided TAP block will be done to the patients using 0.25% bupivacaine, in a dose of (1 ml / kg).
  Arms: group A
Procedure: Caudal Block — ultrasound (US) guided caudal block will be done to the patients using 0.25% bupivacaine, in a dose of (1 ml / kg).
  Arms: group B
Drug: Bupivacaine 0.25% Injectable Solution — Dose 1ml /kg of patient body weight
Device: Ultra-sound guidance — using superficial high frequency probe to guide regional anesthesia

SUMMARY:
The use of pediatric regional anesthesia has increased because of its effective pain control, improved safety profile of local anesthetic agents, in addition to the introduction of ultra-sound. At present, caudal block is one of the most common regional anesthetic techniques employed in pediatric surgery. In addition to providing postoperative analgesia, caudal block significantly reduces intraoperative analgesic requirements and upper airway complications. Transversus abdominis plane (TAP) block involves infiltration of local anesthetics to the plane between the internal oblique and transversus abdominis muscles. Indeed, TAP block offers a hemodynamic stability, appropriate intra-operative analgesia and post surgical analgesia of the abdominal wall.

DETAILED DESCRIPTION:
The use of pediatric regional anesthesia has increased because of its effective pain control, improved safety profile of local anesthetic agents, in addition to the introduction of ultra-sound.

At present, caudal block is one of the most common regional anesthetic techniques employed in pediatric surgery. In addition to providing postoperative analgesia, caudal block significantly reduces intraoperative analgesic requirements and upper airway complications.

However, in recent days there is a trend toward the use of peripheral nerve blockade wherever applicable, given the lower incidences of adverse effects when compared with neuron-axial techniques. Furthermore, there may be specific anatomic variations or abnormalities which preclude the use of caudal block.

The abdominal wall consists of three muscular layers, the external oblique abdominis muscle (EOAM), the internal oblique abdominis muscle (IOAM), and the tranversus abdominis muscle (TAM), and their associated fascial sheaths. The central abdominal wall also includes the rectus abdominis muscles and its associated fascial sheath. This muscular wall is innervated by nerve afferents that course through the transversus abdominis neuron-fascial plane.

Transversus abdominis plane (TAP) block involves infiltration of local anesthetics to the plane between the internal oblique and transversus abdominis muscles. Indeed, TAP block offers a hemodynamic stability, appropriate intra-operative analgesia and post surgical analgesia of the abdominal wall.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American society of anesthiologists) physical status grade I-II.
* Operations not extending more than two hours.
* Unilateral surgeries.

Exclusion Criteria:

* Refusal of parents.
* Urgent cases.
* Bilateral or Complicated hernias (i.e., obstructed, strangulated, irreducible …).
* Other contraindication of regional anesthesia e.g. septic focus at site of injection, patients on anticoagulant therapy or suffering from coagulopathy, allergy to local anesthetic drug.
* Prolonged operations more than two hours.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
Time for first analgesic request | 24 hours after surgery
  by investigator till hospital discharge, then through telephone with parents after discharge

SECONDARY OUTCOMES:
Total Opioid consumpsion | During operation
  Total amount of intra-operative fentanyl consumption.
Total Ibuprofen consumption | 24 hours after surgery
  Total amount of oral ibuprofen consumption postoperative.
post operative pain score. | 2 , 4 , 8 , 12 & 24 hours after surgery.
  Pain assessment by Children's Hospital of Eastern Ontario Pain Scale (CHEOPS) by investigator till hospital discharge, then through telephone with parents after discharge
parents satisfaction score. | 24 hours after surgery
  satisfaction were measured on a 5 point scale of "extremely dissatisfied" to "extremely satisfied" as follows: 1- Completely dissatisfied (worst), 2- Dissatisfied 3- Not satisfied, nor dissatisfied, 4- Satisfied, 5- Completely satisfied (best).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Refky, MD, Study Chair — Faculty of medicine, zagazig university, Egypt; Doaa M Farid, MD, Study Chair — Faculty of medicine, zagazig university, Egypt; Ayat A Amer, MD, Study Director — Faculty of medicine, zagazig university, Egypt
Locations (1):
- Faculty of medicine, Zagazig University., Zagazig, Alsharkia, Egypt